CLINICAL TRIAL: NCT06975007
Title: Comparing the Stress-Reducing Effects of a Robotic Pet and a Weighted Toy: A Randomised Experimental Study
Brief Title: Comparing the Stress-Reducing Effects of a Robotic Pet and a Weighted Toy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Nina Akulova, student, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23002
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Stress
Keywords: Stress reduction; Robotic pet; Paro; Weighted sensory toy; Deep pressure stimulation; Acute stress; Trier Social Stress Test (TSST); Heart rate; Blood pressure; Human-robot interaction; Sensory modulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups: interaction with a robotic companion (Paro), interaction with a weighted sensory toy or a control group with no intervention. Each participant will experience only one intervention condition following the stress induction task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paro Robot Interaction (Experimental): Participants will interact with Paro, a robotic companion seal, for 15 minutes following a stress induction task. Paro responds to touch and sound.
  Interventions: Device: Paro Robotic Companion Seal
- Weighted Toy Interaction (Experimental): Participants will hold and interact with a weighted sensory toy for 15 minutes following a stress induction task. The weighted toy provides deep pressure stimulation for calming effects.
  Interventions: Device: Weighted Sensory Toy
- Control Group (No Intervention) (No Intervention): Participants will sit quietly for 15 minutes without any intervention following a stress induction task. This group allows natural recovery from stress without external aids.

INTERVENTIONS:
Device: Paro Robotic Companion Seal — Paro is an interactive robotic companion designed to simulate the behaviour of a baby harp seal. It responds to touch, light, sound, posture and temperature, providing tactile and social interaction for stress relief.
  Arms: Paro Robot Interaction
Device: Weighted Sensory Toy — A soft, weighted animal-shaped toy (dog) designed to provide deep pressure stimulation. Participants hold or interact with the toy for 15 minutes following a stress induction task to promote relaxation and stress reduction.
  Arms: Weighted Toy Interaction

SUMMARY:
The goal of this trial is to learn whether interacting with a robotic pet (Paro) or holding a weighted sensory toy can reduce stress in healthy adults after an acute stressful experience. The main questions it aims to answer are:

* Does interacting with Paro or holding a weighted toy lower self-reported stress and anxiety levels?
* Does interacting with Paro or holding a weighted toy lower physiological markers of stress, such as heart rate and blood pressure?

Researchers will compare interaction with Paro (robotic pet), interaction with a weighted sensory toy and a control group with no intervention to see which method is most effective in reducing stress.

Participants will:

1. Complete a stress induction task (Trier Social Stress Test);
2. Be randomly assigned to interact with Paro, hold a weighted toy, or sit quietly without intervention;
3. Have their heart rate and blood pressure measured;
4. Complete surveys about their stress, anxiety and mood before and after the intervention.

DETAILED DESCRIPTION:
The study investigates the immediate effectiveness of interacting with an interactive robotic pet (Paro, a robotic seal) or a weighted sensory modulation toy for reducing acute stress and anxiety. It aims to determine the comparative efficacy of these interventions relative to a control condition involving quiet relaxation. Participants will be randomly assigned to one of three experimental conditions: interaction with Paro, interaction with a weighted sensory toy, or a control group with no intervention.

All participants will first complete baseline measurements, including self-reported anxiety and stress assessments using validated instruments (State-Trait Anxiety Inventory, Positive and Negative Affect Schedule, and Visual Analog Scale), as well as physiological indicators of stress (heart rate and blood pressure). Subsequently, participants will undergo the Trier Social Stress Test (TSST), a validated procedure involving a brief public speaking task and mental arithmetic performed under evaluative conditions designed to induce moderate stress. Following the stress induction, participants will repeat stress and anxiety assessments and physiological measurements. They will then engage in their assigned intervention for 15 minutes. Post-intervention measurements of stress and anxiety, physiological markers, and perceived enjoyment/ engagement will be collected. Participants will also provide qualitative feedback regarding their intervention experiences.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* fluent in English
* free from diagnosed anxiety or stress-related disorders

Exclusion Criteria:

* cardiovascular conditions that may affect heart rate and blood pressure measurements
* existing anxiety disorders or panic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in affect (Positive and Negative Affect Schedule - PANAS) | Baseline, immediately after stress induction and immediately after intervention (approximately 1 hour total)
  Positive and negative affect will be assessed using the PANAS at three time points. The primary outcome is the change in both subscale scores from post-stress to post-intervention across groups.
Change in state anxiety scores (STAI-State short form) | Baseline, immediately after stress induction, and immediately after intervention (~1 hour total)
  Participants' state anxiety will be measured at baseline, after the stress induction task, and after the intervention using the six-item short-form State-Trait Anxiety Inventory (STAI-State). The primary comparison will be change in scores from post-stress to post-intervention across the three groups.
Change in subjective stress levels (Visual Analog Scale for stress) | Baseline, immediately after stress induction, and immediately after intervention (~1 hour total)
  Participants will rate their current level of stress on a 100 mm Visual Analog Scale at three time points. The change from post-stress induction to post-intervention will be compared across groups.

SECONDARY OUTCOMES:
Change in heart rate | Baseline, immediately after stress induction and immediately after intervention (approximately 1 hour total)
  Participants' heart rate will be measured at three time points (baseline, post-stress induction and post-intervention) using an automated digital monitor. HR will be measured in beats per minute (BPM).
Change in blood pressure | Baseline, immediately after stress induction and immediately after intervention (approximately 1 hour total)
  Participants' blood pressure will be measured at three time points (baseline, post-stress induction and post-intervention) using an automated digital monitor. BP will be recorded in millimeters of mercury (mmHg), capturing both systolic (SBP) and diastolic (DBP) values.
Participant ratings of enjoyment and engagement (VAS scales) | Immediately after intervention (within approximately 1 hour of study start)
  Participants in the Paro and Weighted Sensory Toy groups will complete visual analog scales (VAS) rating their enjoyment and engagement with the intervention. Each scale is 100 mm in length, anchored with "Not at all" (0 mm) to "Extremely" (100 mm). Higher scores indicate greater enjoyment or engagement.
Qualitative feedback on participant experience | Immediately after intervention (within approximately 1 hour of study start)
  Participants will provide open-ended qualitative feedback about their experience with their assigned intervention (Paro, Weighted Toy or Control). Responses will be analysed using thematic analysis to identify common themes.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Broadbent, Professor, Principal Investigator — Department of Psychological Medicine, The University of Auckland
Locations (1):
- University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
confidential. Ethical requirements are to keep individual data confidential.